CLINICAL TRIAL: NCT03229408
Title: Treating Inflammation in Polycystic Ovary Syndrome to Ameliorate Ovarian Dysfunction
Acronym: TIN-PCOS-AOD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Frank Gonzalez, Director, Laboratory for Reproductive Endocrine and Inflammation Research, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2017-0476; R01DK107605 (NIH)
Record Dates: First submitted 2017-07-15; First posted 2017-07-25 (Actual); Results first posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-05

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Inflammation; Hyperandrogenism; Anovulation; Insulin Resistance
MeSH Terms: conditions — Polycystic Ovary Syndrome; Inflammation; Hyperandrogenism; Anovulation; Insulin Resistance | interventions — salicylsalicylic acid; Sodium Salicylate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Salsalate-Treated Lean PCOS without IR (Experimental): n=15
  Interventions: Drug: Salsalate
- Placebo-Treated Lean PCOS without IR (Placebo Comparator): n=15
  Interventions: Other: Placebo
- Salsalate-Treated Lean PCOS with IR (Experimental): n=15
  Interventions: Drug: Salsalate
- Placebo-Treated Lean PCOS with IR (Placebo Comparator): n=15
  Interventions: Other: Placebo
- Salsalate-Treated Obese PCOS (Experimental): n=15
  Interventions: Drug: Salsalate
- Placebo-Treated Obese PCOS (Placebo Comparator): n=15
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Salsalate — Lean PCOS Arms: Salsalate 1.5 gm PO bid; Obese PCOS Arm: Salsalate 2.0 gm PO bid
  Other Names: Disalcid®; Salsitab®; Amigesic®
  Arms: Salsalate-Treated Lean PCOS with IR; Salsalate-Treated Lean PCOS without IR; Salsalate-Treated Obese PCOS
Other: Placebo — Appears identical to experimental drug
  Arms: Placebo-Treated Lean PCOS with IR; Placebo-Treated Lean PCOS without IR; Placebo-Treated Obese PCOS

SUMMARY:
Polycystic Ovary Syndrome (PCOS) is characterized by hyperandrogenism, ovulatory dysfunction and polycystic ovaries. Insulin resistance (IR) is a common feature of PCOS, and the resultant hyperinsulinemia is theorized to promote hyperandrogenism in the disorder. However, 30-50% of women with PCOS who are lean do not have insulin resistance. Women with PCOS also exhibit chronic low-grade inflammation. In PCOS, glucose ingestion activates nuclear factor ĸB (NFĸB), the cardinal signal of inflammation culminating in upregulation of the inflammation pathway within mononuclear cells (MNC). This phenomenon is independent of excess adiposity and is highly correlated with circulating androgens. In addition, in vitro exposure to proinflammatory stimuli is capable of directly stimulating ovarian theca cell androgen production. Nonacetylated salicylates suppress NFĸB activation and are well tolerated in humans.

The proposed research is a randomized double-blind placebo-controlled study of 90 women with PCOS. Forty-five subjects with PCOS (15 lean without IR), 15 lean with IR and 15 obese) receiving salsalate, a nonacetylated salicylate, at an oral dose of 3-4 gm daily for 12 weeks will be compared with 45 age- and body-composition-matched control women with PCOS receiving placebo. The overarching hypothesis is that inflammation contributes to ovarian dysfunction, independent of excess adiposity or IR.

The specific aims are, I: To examine the effect of salsalate administration on the ovarian capacity to secrete androgen and on insulin sensitivity in PCOS. II: To examine the effect of salsalate administration on the inflammatory response of mononuclear cells induced by lipid ingestion and glucose infusion in PCOS. The approach involves evaluation of ovarian androgen secretion in response to human chorionic gonadotropin (HCG) administration and insulin sensitivity during the euglycemic phase of a two-step pancreatic clamp along with ovulation monitoring before and after salsalate administration. The inflammatory response of MNC to lipid ingestion and the hyperglycemic phase of the two-step clamp will also be evaluated during treatment by measuring reactive oxygen species, the mRNA and protein content of inflammation markers, NFĸB activation and cytokine release in culture.

The investigators expect that women with PCOS receiving salsalate will exhibit decreased ovarian androgen secretion and reduced inflammation regardless of adiposity or IR status. These results will be significant if they show a causal contribution of inflammation to ovarian dysfunction in PCOS, thus improving our understanding of the pathogenesis of PCOS, opening previously unexplored therapeutic avenues that are not necessarily dependent on improving IR, and guiding the design of future studies aimed at determining what interventions will optimally attenuate inflammation in PCOS to reduce medical disease and enhance fertility.

DETAILED DESCRIPTION:
PCOS is characterized by hyperandrogenism, ovarian dysfunction and polycystic ovarian morphology. Obesity and IR are common features of PCOS. Under the current model of pathophysiology of PCOS, the compensatory hyperinsulinemia of IR is the primary driver of hyperandrogenism. This concept was born from the cross-sectional observation that insulin is positively correlated with androgens in obese women with PCOS, and is supported by reports of increased androgen production from theca cells obtained from obese women with PCOS following insulin exposure in vitro and increases in circulating androgens in women with PCOS following insulin infusion in vivo. However, these in vitro - in vivo responses were elicited with supraphysiological insulin concentrations. Physiological insulin infusion on the other hand does not augment androgen levels in PCOS. The current model also does not explain the cause of hyperandrogenism and ovarian dysfunction in the 30-50% of women with PCOS who are lean and lack IR. Thus, some other factor contributes to these abnormalities in PCOS.

The investigators have shown that ingestion of glucose and saturated fat elicits an inflammatory response from circulating MNC in lean women with PCOS who lack excess abdominal adiposity. The hallmark of this response is increased activation of NFĸB, the cardinal signal of inflammation. These findings illustrate the separate and discrete role of MNC in manifesting inflammation in PCOS and that MNC are an excellent model to assess systemic inflammation in PCOS.

The investigators have also shown that in PCOS, there is a link between molecular markers of inflammation from MNC and circulating androgens. Chronic suppression of ovarian androgen production does not ameliorate inflammation in lean women with PCOS. However, in vitro exposure of ovarian theca cells to proinflammatory stimuli upregulates CYP17, the androgen producing enzyme and increases testosterone.

Salsalate is an inexpensive, safe, well-tolerated, well-understood anti-inflammatory agent that inhibits NFĸB activation when used at higher doses. The salsalate dose required to achieve a salicylate level in the upper therapeutic range is dependent on body mass. This is achieved in lean individuals using 3.0 gm/day as the maximum dose recommended in the salsalate package insert. Individuals across the obese range (30-40 kg/m2) require >3.0 gm/day to achieve the same objective. Salsalate and other salicylates have also been shown to decrease IR. However, the ability of salsalate to decrease IR would not be necessary if the beneficial anti-inflammatory effect of salsalate to reduce hyperandrogenism is on the ovaries. In fact, we have shown that in lean insulin-sensitive women with PCOS, salsalate reduces HCG-stimulated ovarian androgen secretion by 44% and normalizes basal testosterone levels. Studies performed by the investigators in MNC also confirm the ability of salsalate to suppress NFĸB activation. Together these observations validate the use of these measurements as endpoints to assess the effects of salsalate to probe the pathophysiology of PCOS.

Salsalate raises circulating insulin due to its ability to decreased insulin clearance from the liver which confounds the assessment of insulin sensitivity from post-treatment hyperinsulinemic-euglycemic clamp studies. Performance of a novel minimal model-based analysis from an insulin-modified frequently-sampled intravenous glucose tolerance test (FS-IVGTT) is able to address this confounding factor. With this approach, hepatic and extrahepatic insulin clearance can be estimated before and after salsalate treatment to obtain measures of insulin sensitivity that take into account the salsalate-induced alteration in insulin clearance.

In this context, the rationale for the proposed study revolves around the concept that in PCOS, inflammation contributes to ovarian dysfunction independent of excess adiposity or IR, and may also improve insulin sensitivity when IR is present. The investigators will undertake a 12-week randomized, double-blind, placebo-controlled trial to test the link between inflammation and ovarian androgen secretion in PCOS unrelated to IR. If this study of pathophysiology demonstrates beneficial effects, this will pave the way for developing novel therapies for ovarian dysfunction in PCOS.

The main objective of this proposal is to evaluate the ability of salsalate to reduce ovarian androgen secretion, induce ovulation and decrease lipid-stimulated inflammation independent of body composition and IR in women with PCOS; and to also improve insulin sensitivity in IR women with PCOS. Effects of salsalate will be assessed based on the following aims:

Specific Aim 1. To examine the effects of salsalate administration on the ovarian capacity to secrete androgens, menstrual function, and insulin sensitivity in PCOS.

The hypothesis for this aim is that salsalate treatment will decrease HCG-stimulated ovarian androgen secretion and induce ovulation in women with PCOS regardless of body composition or IR status; and may also improve insulin sensitivity in IR women with PCOS. The investigators will test this hypothesis in a randomized double-blind placebo-controlled study. The ovarian androgen response to HCG administration will be evaluated in women with PCOS (15 lean with IR, 15 lean without IR and 15 obese) before and after administration of a therapeutic salsalate dose for ~12 weeks compared with women with PCOS receiving placebo for ~12 weeks (15 lean with IR, 15 lean without IR and 15 obese). Ovulation monitoring and assessment of insulin sensitivity during FS-IVGTT will be performed before and after salsalate or placebo administration. It is anticipated that salsalate will reduce HCG-stimulated ovarian androgen secretion, induce ovulation regardless of body composition or IR status when compared with placebo. It is also anticipated that salsalate will increase insulin sensitivity in IR women with PCOS compared with placebo.

Specific Aim 2. To examine the effect of salsalate administration on the inflammatory response of mononuclear cells induced by lipid ingestion in PCOS.

The hypothesis for this aim is that salsalate administration will down-regulate inflammatory signal transduction and cytokine production within MNC following lipid ingestion in women with PCOS regardless of body composition or IR status. The investigators will test this hypothesis using the study design described in Aim 1. The inflammatory response of MNC to a cream challenge test will be evaluated in women with PCOS before and after salsalate treatment. It is anticipated that lipid-induced inflammation will decrease with salsalate use regardless of body composition or IR status when compared with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PCOS based on the presence of hyperandrogenism (skin manifestations of androgen excess such as hirsutism, acne or temporal balding - or -elevation of at least one serum androgen [i.e. total testosterone, free testosterone, androstenedione or dehydroepiandrosterone-sulphate] using predetermined local laboratory cutoffs), oligo/amenorrhea and evidence of withdrawal bleeding after progestin administration.
* 18-40 years of age.
* Good health as evidenced by medical history, physical examination and gynecologic examination within 30 days prior to starting the study.
* Willingness to provide informed consent according to the guidelines of the University of Illinois at Chicago (UIC) Institutional Review Board (IRB).
* Willingness to use double-barrier contraception such as condoms and topical spermicide (foam, cream or gel), condom and diaphragm, diaphragm and topical spermicide or sponge with topical spermicide if sexually active. Use of a non-hormonal intrauterine device (IUD), or permanent sterilization of the subject or her partner (i.e. tubal ligation or vasectomy) is also acceptable in all instances.

Exclusion Criteria:

* Hyperprolactinemia.
* Uncontrolled thyroid disease.
* Evidence of Cushing's syndrome, nonclassic congenital adrenal hyperplasia or a hormone producing tumor based on physical findings and serum androgen levels on initial screening.
* Known or suspected pregnancy.
* Regular vigorous physical activity during previous 6 months.
* Use of any medications known to affect carbohydrate or sex hormone metabolism such as oral contraceptives, progestins, glucocorticoids or insulin sensitizing agents within 30 days of beginning the study.
* Acute or chronic inflammatory illnesses (e.g. upper respiratory infection, asthma, rheumatoid arthritis or systemic lupus erythematosus).
* Type 1 or type 2 diabetes mellitus defined as having a fasting glucose >126 mg/dl and/or a 2-hour postprandial glucose >200 mg/dl.
* Regular smoking defined as more than 2 cigarettes a month, or any smoking within 30 days of beginning the study.
* History of any illness exacerbated by salicylate use (e.g. peptic ulcer hepatic or renal disease, anemia, thrombosis, coagulopathy, congestive heart failure, hypertension or gout).
* Allergy to salicylate or dairy products.
* Medication use interacting with salicylates such as anti-platelet drugs (e.g. cilostazol, clopidogrel), anticoagulants (e.g. enoxaparin, heparin, warfarin), corticosteroids (e.g., prednisone), certain diabetes drugs (e.g. sulfonylureas such as glyburide), certain anti-seizure drugs (e.g. phenytoin, valproic acid), cidofovir, cyclosporine, drugs for gout (e.g. probenecid, sulfinpyrazone), anti-hypertensives (e.g. angiotensin converting enzyme inhibitors such as captopril, angiotensin II receptor antagonists such as losartan, and beta blockers such as metoprolol), drugs that affect the acidity of urine (e.g. ammonium chloride, acetazolamide), lithium, methotrexate, oral bisphosphonates (e.g. alendronate), pemetrexed, selective serotonin reuptake inhibitor antidepressants (e.g. fluoxetine, sertraline), tenofovir, and diuretics (furosemide, hydrochlorothiazide, spironolactone).

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Polycystic ovary syndrome is a female endocrine disorder.
Enrollment: 60 (Actual)
Dates: Start 2018-12-05 (Actual); Primary Completion 2024-02-14 (Actual); Study Completion 2024-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank González, M.D., Principal Investigator — University of Illinois at Chicago
Locations (1):
- Frank González, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gonzalez F, Mather KJ, Considine RV, Abdelhadi OA, Acton AJ. Salicylate administration suppresses the inflammatory response to nutrients and improves ovarian function in polycystic ovary syndrome. Am J Physiol Endocrinol Metab. 2020 Oct 1;319(4):E744-E752. doi: 10.1152/ajpendo.00228.2020. Epub 2020 Aug 24. PMID 32830548
- See also: Principal Investigator's research laboratory and research program description — https://chicago.medicine.uic.edu/departments/academic-departments/obstetrics-and-gynecology/laboratory-for-reproductive-endocrine-and-inflammation-research/
- See also: Principal Investigator's National Center for Biotechnology Information MyBibliography — https://www.ncbi.nlm.nih.gov/myncbi/browse/collection/41157534/?sort=date&direction=descending
- See also: Principal Investigator's research profile — https://www.researchgate.net/profile/Frank-Gonzalez-7
- See also: Principal Investigator's career profile — https://www.doximity.com/pub/frank-gonzalez-md

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 60 volunteers enrolled, 35 of them never entered the protocol for the following reasons: Lost to follow up before screening completed during intermittent COVID-19 person-to-person human research suspensions (n=21); Declined study participation despite eligibility after screening (n=6); Ineligible after screening (n=8). The remaining 25 volunteers were entered into the study protocol.
Groups:
- Experimental: Salsalate-Treated PCOS: Lean PCOS (BMI 18.0-24.9 kg/m2): Salsalate 1.5 gm PO bid or Obese PCOS (BMI 30.0-39.9 kg/m2): Salsalate 2.0 gm PO bid
- Placebo Comparator: Placebo-Treated PCOS: Lean PCOS (BMI 18.0-24.9 kg/m2) or Obese PCOS (BMI 30.0-39.9 kg/m2): Placebo appears identical to experimental drug
Period: Overall Study
Arm/Group | Experimental: Salsalate-Treated PCOS | Placebo Comparator: Placebo-Treated PCOS
Started | 14 | 11
Completed | 6 | 7
Not Completed | 8 | 4
Not completed — Withdrawal by Subject | 4 | 1
Not completed — Adverse Event | 2 | 0
Not completed — Pregnancy | 0 | 1
Not completed — Required to stopped during intermittent COVID-19 person-to-person human research suspensions | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental: Salsalate-Treated PCOS | Placebo Comparator: Placebo-Treated PCOS | Total
Number analyzed (Participants) | 14 | 11 | 25
Age, Continuous [Mean (Standard Deviation); unit: Years] | 28 (4) | 29 (4) | 28 (4)
Sex: Female, Male [Count of Participants; unit: Participants] — Only females participated in the study
  Participants
    Female | 14 | 11 | 25
    Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 4 | 11
  Not Hispanic or Latino | 7 | 7 | 14
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 5 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 3 | 1 | 4
  More than one race | 7 | 4 | 11
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: Participants]
  United States | 14 | 11 | 25
Body Mass Index [Mean (Standard Deviation); unit: Kilos Per Meters Squared (kg/m2)] | 31.3 (5.9) | 28.5 (6.4) | 30.0 (6.2)
Total Body Fat [Mean (Standard Deviation); unit: Cubic Centimeters (cm3)] — Body composition assessment by magnetic resonance imaging Population: Only 13 participants assigned to the Experimental: Salsalate-Treated PCOS arm underwent magnetic resonance imaging. One (1) participant assigned to the Experimental: Salsalate-Treated PCOS arm who did not complete the study did not undergo magnetic resonance imaging due to the contradiction of having a copper intrauterine conception device in situ.
  Cubic Centimeters (cm3)
    number analyzed (Participants) | 13 | 11 | 24
    (all) | 21981 (5086) | 18273 (6720) | 20282 (6057)
Total Abdominal Fat [Mean (Standard Deviation); unit: Cubic Centimeters (cm3)] — Body composition assessment by magnetic resonance imaging Population: Only 13 participants assigned to the Experimental: Salsalate-Treated PCOS arm underwent magnetic resonance imaging. One (1) participant assigned to the Experimental: Salsalate-Treated PCOS arm who did not complete the study did not undergo magnetic resonance imaging due to the contradiction of having a copper intrauterine conception device in situ.
  Cubic Centimeters (cm3)
    number analyzed (Participants) | 13 | 11 | 24
    (all) | 13710 (4741) | 11867 (5322) | 12865 (4992)
Visceral Fat [Mean (Standard Deviation); unit: Cubic Centimeters (cm3)] — Body composition assessment by magnetic resonance imaging Population: Only 13 participants assigned to the Experimental: Salsalate-Treated PCOS arm underwent magnetic resonance imaging. One (1) participant assigned to the Experimental: Salsalate-Treated PCOS arm who did not complete the study did not undergo magnetic resonance imaging due to the contradiction of having a copper intrauterine conception device in situ.
  Cubic Centimeters (cm3)
    number analyzed (Participants) | 13 | 11 | 24
    (all) | 3817 (1390) | 4487 (5439) | 4125 (3740)
Basal Testosterone Level [Mean (Standard Deviation); unit: Nanograms per Deciliter (ng/dL)] — Serum measurement by chemiluminescence (Siemens Immulite 2000, Cary, NC)
  Nanograms per Deciliter (ng/dL) | 70 (9) | 67 (6) | 69 (8)
Basal Androstenedione Level [Mean (Standard Deviation); unit: Nanograms per Milliliter (ng/mL)] — Serum measurement by ELISA (ALPCO Diagnostics, Salem, NH)
  Nanograms per Milliliter (ng/mL) | 3.85 (0.53) | 3.66 (0.46) | 3.77 (0.50)
HCG-stimulated Testosterone Area Under the Curve [Mean (Standard Deviation); unit: Nanograms*Hour per Deciliter (ng*hr/dL)] — Data was generated from the pre-treatment HCG stimulation test. Area under the curve calculated for serum measurements by chemiluminescence (Siemens Immulite 2000, Cary, NC) from blood samples drawn 0, 24, 48 and 72 hours after HCG administration.
  Nanograms*Hour per Deciliter (ng*hr/dL) | 7830 (1208) | 7673 (1109) | 7761 (1145)
HCG-stimulated Androstenedione Area Under the Curve [Mean (Standard Deviation); unit: Nanograms*Hour per Milliliter (ng*hr/mL)] — Data was generated from the pre-treatment HCG stimulation test. Area under the curve calculated for serum measurements by ELISA (ALPCO Diagnostics, Salem, NH) from blood samples drawn 0, 24, 48 and 72 hours after HCG administration.
  Nanograms*Hour per Milliliter (ng*hr/mL) | 422 (69) | 415 (40) | 419 (57)
Insulin Sensitivity (SI) [Mean (Standard Deviation); unit: Microunits/Milliliter/Minute (µU/mL/min)] — Data was generated from the pre-treatment frequently-sampled intravenous glucose tolerance test (FS-IVGTT). Calculated using the Bergman minimal model (Am J Physiol 1979, 236:E667-E677) from serum insulin measurements using blood samples drawn while fasting at -20, -10, -1, 0, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 14, 16, 19, 22, 23, 24, 25, 27, 30, 40, 50, 60, 70, 80, 90, 100, 120, 150, 180 and 240 minutes. Population: Although 25 participants entered the protocol, baseline measures of insulin sensitivity are only provided for the 13 participants (6 salsalate arm; 7 placebo arm) with both pre- and post- treatment samples. Due to cost, pre-treatment samples from the 12 participants (8 salsalate arm; 4 placebo arm) without post-treatment samples to generate outcome data were not analyzed since this would not yield meaningful results to address the study aims, and there is no plan to analyze these in the future.
  Microunits/Milliliter/Minute (µU/mL/min)
    number analyzed (Participants) | 6 | 7 | 13
    (all) | 2.86 (0.76) | 3.50 (0.63) | 3.20 (0.74)
Lipid-stimulated ROS Generation [Mean (Standard Deviation); unit: Percent Change] — Data was generated from the pre-treatment cream challenge test. Measured by chemiluminescence in mononuclear cells isolated from blood samples drawn while fasting (0 hour) and 2 hours after cream ingestion. Percent change was calculated using the 2 hour ROS value (mV) minus the 0 hour ROS value (mV) divided by the 0 hour ROS value (mV), multiplied by 100.
  Percent Change | 122 (43) | 102 (41) | 114 (42)
Lipid-stimulated NFкB Activation [Mean (Standard Deviation); unit: Percent Change] — Data was generated from the pre-treatment cream challenge test. Quantified in nuclear extracts by oligonucleotide-based ELISA (Active Motif, Carlsbad, CA) in mononuclear cells isolated from blood samples drawn while fasting (0 hour) and 2 hours after cream ingestion. Percent change was calculated using the 2 hour NFкB band intensity value determined by densitometry minus the 0 hour NFкB band intensity value divided by the 0 hour NFкB band intensity value, multiplied by 100.
  Percent Change | 93 (35) | 134 (84) | 111 (64)
Lipid-stimulated TNFα Secretion [Mean (Standard Deviation); unit: Picograms per Milliliter (pg/mL)] — Data was generated from the pre-treatment cream challenge test. Measured in culture supernatants by ELISA (Quantikine, R&D Systems, Minneapolis, MN) in mononuclear cells isolated from blood samples drawn while fasting (0 hour) and 2 hours after cream ingestion. Absolute change was calculated using the 2 hour TNFα value (pg/mL) minus the 0 hour TNFα value (pg/mL).
  Picograms per Milliliter (pg/mL) | 13.1 (7.0) | 14.0 (3.3) | 13.5 (5.6)

OUTCOME MEASURES:

1. Primary Outcome: Aim 1: HCG-stimulated Testosterone Area Under the Curve
Description: Data was generated from the post-treatment HCG stimulation test. Area under the curve calculated for serum measurements by chemiluminescence (Siemens Immulite 2000, Cary, NC) from blood samples drawn 0, 24, 48 and 72 hours after HCG administration.
Time Frame: After 12 weeks of salsalate administration
Population: Only 13 of the 25 participants who entered the protocol completed the study consisting of 6 participants assigned to the Experimental: Salsalate-Treated PCOS arm and 7 participants assigned to the Placebo Comparator: Placebo-Treated PCOS arm. The remaining 12 participants did not complete the study consisting of 8 participants assigned to the Experimental: Salsalate-Treated PCOS arm and 4 participants assigned to the Placebo Comparator: Placebo-Treated PCOS arm.
Measure: Mean (Standard Error); unit: Nonograms*Hour per Deciliter (ng*hr/dL)
Arm/Group | Experimental: Salsalate-Treated PCOS | Placebo Comparator: Placebo-Treated PCOS
Number analyzed (Participants) | 6 | 7
Nonograms*Hour per Deciliter (ng*hr/dL) | 4458 (717) | 7775 (539)
Statistical Analysis 1: Comparison: Experimental: Salsalate-Treated PCOS vs Placebo Comparator: Placebo-Treated PCOS; Test type: Superiority; p < 0.004, Unpaired t-test, 2-Sided

2. Primary Outcome: Aim 2: Lipid-stimulated NFкB Activation
Description: Data was generated from the post-treatment cream challenge test. Quantified in nuclear extracts by oligonucleotide-based ELISA (Active Motif, Carlsbad, CA) in mononuclear cells isolated from blood samples drawn while fasting (0 hour) and 2 hours after cream ingestion. Percent change was calculated using the 2 hour NFкB band intensity value determined by densitometry minus the 0 hour NFкB band intensity value divided by the 0 hour NFкB band intensity value, multiplied by 100.
Time Frame: After 12 weeks of salsalate or placebo administration
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Percent Change
Arm/Group | Experimental: Salsalate-Treated PCOS | Placebo Comparator: Placebo-Treated PCOS
Number analyzed (Participants) | 6 | 7
Percent Change | 37 (7) | 89 (17)
Statistical Analysis 1: Comparison: Experimental: Salsalate-Treated PCOS vs Placebo Comparator: Placebo-Treated PCOS; Test type: Superiority; p < 0.03, Unpaired T-test, 2-Sided

3. Secondary Outcome: Aim 1: Insulin Sensitivity (SI)
Description: Data was generated from the post-treatment frequently-sampled intravenous glucose tolerance test (FS-IVGTT). Calculated using the Bergman minimal model (Am J Physiol 1979, 236:E667-E677) from serum insulin measurements using blood samples drawn while fasting at -20, -10, -1, 0, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 14, 16, 19, 22, 23, 24, 25, 27, 30, 40, 50, 60, 70, 80, 90, 100, 120, 150, 180 and 240 minutes.
Time Frame: After 12 weeks of salsalate or placebo adminitration
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Microunits/Milliliter/Minute (µU/mL/min)
Arm/Group | Experimental: Salsalate-Treated PCOS | Placebo Comparator: Placebo-Treated PCOS
Number analyzed (Participants) | 6 | 7
Microunits/Milliliter/Minute (µU/mL/min) | 2.63 (0.43) | 3.71 (0.61)
Statistical Analysis 1: Comparison: Experimental: Salsalate-Treated PCOS vs Placebo Comparator: Placebo-Treated PCOS; Test type: Superiority; p = 0.180, Unpaired t-test, 2-Sided

4. Secondary Outcome: Aim 1: Basal Testosterone Level
Description: Serum measurement by chemiluminescence (Siemens Immulite 2000, Cary, NC).
Time Frame: After 12 weeks of salsalate or placebo administration
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Nanograms per Deciliter (ng/dL)
Arm/Group | Experimental: Salsalate-Treated PCOS | Placebo Comparator: Placebo-Treated PCOS
Number analyzed (Participants) | 6 | 7
Nanograms per Deciliter (ng/dL) | 38 (6) | 67 (3)
Statistical Analysis 1: Comparison: Experimental: Salsalate-Treated PCOS vs Placebo Comparator: Placebo-Treated PCOS; Test type: Superiority; p < 0.002, Unpaired T-test, 2-Sided

5. Secondary Outcome: Aim 1: Basal Androstenedione Level
Description: Serum measurement by ELISA (ALPCO Diagnostics, Salem, NH)
Time Frame: After 12 weeks of salsalate or placebo administration
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Nanograms per Milliliter (ng/mL)
Arm/Group | Experimental: Salsalate-Treated PCOS | Placebo Comparator: Placebo-Treated PCOS
Number analyzed (Participants) | 6 | 7
Nanograms per Milliliter (ng/mL) | 2.42 (0.54) | 3.69 (0.15)
Statistical Analysis 1: Comparison: Experimental: Salsalate-Treated PCOS vs Placebo Comparator: Placebo-Treated PCOS; Test type: Superiority; p < 0.04, Unpaired t-test, 2-Sided

6. Secondary Outcome: Aim 1: HCG-stimulated Androstenedione Area Under the Curve
Description: Data was generated from the post-treatment HCG stimulation test. Area under the curve calculated for serum measurements by ELISA (ALPCO Diagnostics, Salem, NH) from blood samples drawn 0, 24, 48 and 72 hours after HCG administration.
Time Frame: After 12 weeks of salsalate or placebo administration
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Nanograms*Hour per Milliliter (ng*hr/mL)
Arm/Group | Experimental: Salsalate-Treated PCOS | Placebo Comparator: Placebo-Treated PCOS
Number analyzed (Participants) | 6 | 7
Nanograms*Hour per Milliliter (ng*hr/mL) | 224 (24) | 405 (39)
Statistical Analysis 1: Comparison: Experimental: Salsalate-Treated PCOS vs Placebo Comparator: Placebo-Treated PCOS; Test type: Superiority; p < 0.003, Unpaired t-test, 2-Sided

7. Secondary Outcome: Aim 2: Lipid Stimulated ROS Generation
Description: Data was generated from the post-treatment cream challenge test. Measured by chemiluminescence in mononuclear cells isolated from blood samples drawn while fasting (0 hour) and 2 hours after cream ingestion. Percent change was calculated using the 2 hour ROS value (mV) minus the 0 hour ROS value (mV) divided by the 0 hour ROS value (mV), multiplied by 100.
Time Frame: After 12 weeks of salsalate or placebo administration
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Percent Change
Arm/Group | Experimental: Salsalate-Treated PCOS | Placebo Comparator: Placebo-Treated PCOS
Number analyzed (Participants) | 6 | 7
Percent Change | 31 (8) | 95 (8)
Statistical Analysis 1: Comparison: Experimental: Salsalate-Treated PCOS vs Placebo Comparator: Placebo-Treated PCOS; Test type: Superiority; p < 0.0004, Unpaired t-test, 2-Sided

8. Secondary Outcome: Aim 2: Lipid-stimulated TNFα Secretion
Description: Data was generated from the post-treatment cream challenge test. Measured in culture supernatants by ELISA (Quantikine, R&D Systems, Minneapolis, MN) in mononuclear cells isolated from blood samples drawn while fasting (0 hour) and 2 hours after cream ingestion. Absolute change was calculated using the 2 hour TNFα value (pg/mL) minus the 0 hour TNFα value (pg/mL).
Time Frame: After 12 weeks of salsalate or placebo administration
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Picograms per Milliliter (pg/mL)
Arm/Group | Experimental: Salsalate-Treated PCOS | Placebo Comparator: Placebo-Treated PCOS
Number analyzed (Participants) | 6 | 7
Picograms per Milliliter (pg/mL) | 7.9 (1.3) | 15.1 (1.6)
Statistical Analysis 1: Comparison: Experimental: Salsalate-Treated PCOS vs Placebo Comparator: Placebo-Treated PCOS; Test type: Superiority; p < 0.007, Unpaired t-test, 2-Sided

ADVERSE EVENTS:
Time Frame: up to 16 weeks
Arm/Group | Experimental: Salsalate-Treated PCOS | Placebo Comparator: Placebo-Treated PCOS
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/11
Serious Adverse Events (participants affected / at risk) | 1/14 | 0/11
Other Adverse Events (participants affected / at risk) | 1/14 | 0/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: Salsalate-Treated PCOS (N=14) | Placebo Comparator: Placebo-Treated PCOS (N=11)
Drug Reaction with Eosinophilia and Systemic Symptoms (DRESS) Syndrome (Immune system disorders) | 1 (1) | 0 (0) — DRESS Syndrome is a rare delayed allergic response. Fever and body rash began 6½ weeks after starting salsalate. Pulmonary edema ensued requiring intubation for 12 hours. The participant improved dramatically after intravenous steroid therapy.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: Salsalate-Treated PCOS (N=14) | Placebo Comparator: Placebo-Treated PCOS (N=11)
Medication Allergy - Urticaria (Immune system disorders) | 1 (1) | 0 (0) — A pruritic rash on all four extremities and neck consistent with urticaria began 3 days after starting salsalate prompting discontinuation. The rash completely resolved within 10 days after stopping salsalate use.

LIMITATIONS AND CAVEATS:
The COVID-19 pandemic severely stunted participant accrual culminating in a limited sample size of completed subjects (salsalate; n=6; placebo; n=7). Therefore, combining weight class groups was a reasonable approach to compare outcome measures in salsalate versus placebo.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-09): https://cdn.clinicaltrials.gov/large-docs/08/NCT03229408/Prot_SAP_000.pdf